CLINICAL TRIAL: NCT07345663
Title: Modified Continuous Versus Interrupted Choledochotomy Closure in LCBDE With T-Tube Drainage: A Propensity Score-Matched Cohort Study
Brief Title: Modified Continuous Versus Interrupted Choledochotomy Closure in LCBDE With T-Tube Drainage
Status: Completed | Type: Observational
Sponsor: Yantai Affiliated Hospital of Binzhou Medical University (Other)
Responsible Party: Principal Investigator, Piyou Ji, associate chief physician, Yantai Affiliated Hospital of Binzhou Medical University
Other Study IDs: LW-202601; F-KY-0022-20220325-01 (Other: Yantai affiliated hospital of Binzhou Medical University)
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Common Bile Duct Calculi
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Modified Continuous Suturing
  Interventions: Procedure: Modified continuous suture
- Interrupted Suturing
  Interventions: Procedure: Interrupted suture

INTERVENTIONS:
Procedure: Modified continuous suture — Modified continuous suture was performed using 4-0 knotless barbed polydioxanone sutures (Quill™, Surgical Specialties Corporation). A continuous full-thickness suture was placed from the distal (duodenal) end to the proximal (hepatic) end, with bites of approximately 2 mm and a stitch interval of 3-4 mm. After completion of the continuous closure, 1-2 reinforcing stitches were placed in the opposite direction (from proximal to distal), and the suture was secured by tying to the tail end of the initial stitch.
  Groups: Modified Continuous Suturing
Procedure: Interrupted suture — Interrupted suture was performed using 4-0 antibacterial monofilament polydioxanone sutures (PDS™ Plus, Ethicon, LLC). Interrupted sutures were placed from the distal (duodenal) end to the proximal (hepatic) end, with bites of approximately 2 mm and a stitch interval of 3-4 mm; each stitch was tied separately. An additional 1-2 reinforcing stitches (transverse or figure-of-eight) were placed around the T-tube exit site to enhance apposition between the choledochotomy edge and the tube wall.
  Groups: Interrupted Suturing

SUMMARY:
This observational study aims to compare two techniques for closing the common bile duct incision (choledochotomy) after laparoscopic common bile duct exploration (LCBDE) with T-tube drainage. Interrupted suturing is commonly used, but it can be time-consuming during laparoscopic surgery. A modified continuous suturing approach may improve efficiency while maintaining safety.

We will retrospectively review patients who underwent LCBDE with T-tube drainage at our institution. Patients will be grouped according to the choledochotomy closure technique used during routine clinical care (modified continuous suturing versus conventional interrupted closure). To reduce baseline differences between groups, propensity score matching based on preoperative and intraoperative characteristics will be applied.

The primary outcome is choledochotomy closure time. Secondary outcomes include total operative time and perioperative safety outcomes, such as bile leakage and other postoperative complications, as well as short-term postoperative recovery indicators. This study will provide comparative evidence on operative efficiency and safety of continuous versus interrupted choledochotomy closure in the setting of LCBDE with T-tube drainage.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≥18 years; (2) imaging-confirmed CBDS; (3) intraoperative placement of a T-tube; and (4) Common bile duct (CBD) diameter ≥6 mm

Exclusion Criteria:

* coagulopathy, severe cognitive impairment, multiple intrahepatic stones, biliary stricture, malignancy, liver cirrhosis, severe acute pancreatitis (BISAP score ≥3), and acute cholangitis complicated by septic shock, classified as Grade III according to the Tokyo Guidelines 2018

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who underwent laparoscopic common bile duct exploration (LCBDE) with T-tube drainage at our institution between January 2020 and November 2024. Inclusion criteria include patients who had choledochotomy closure performed with either modified continuous suturing (MCS) or interrupted suturing (IS). Patients were retrospectively reviewed, and baseline characteristics such as age, gender, stone burden, and ASA classification were collected. Exclusion criteria include patients with incomplete data or those who underwent procedures other than LCBDE.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Choledochotomy Closure Time | Closure time is measured intraoperatively during the procedure and recorded once closure is complete.
  The time taken to complete choledochotomy closure, from the beginning of suturing to the completion of the final knot. This measure is recorded in minutes for each patient.

SECONDARY OUTCOMES:
Total Operative Time | The total operative time is measured during the procedure, from the first incision to the final closure.
  The total time from the initiation of the procedure to the completion of the surgery. This includes all steps of the surgery, from incision to closure.

OTHER OUTCOMES:
Intraoperative Blood Loss | Blood loss is recorded intraoperatively at the end of the surgery, based on visual estimation and suction collection.
  The total estimated blood loss during the surgery, as measured by the surgeon and recorded at the end of the procedure. This is typically recorded in milliliters.

CONTACTS AND LOCATIONS:
Locations (1):
- Yantai affiliated hospital of Binzhou Medical University, Yantai, Shandong, China